CLINICAL TRIAL: NCT01616875
Title: A Phase II Trial of Combination Cabazitaxel and Cisplatin Chemotherapy in the Neo-adjuvant Treatment of Transitional Cell Carcinoma of the Urinary Bladder
Brief Title: Bristol Bladder Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospitals Bristol and Weston NHS Foundation Trust (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ON/2011/3775; 2011-004090-82 (EudraCT Number)
Record Dates: First submitted 2012-05-17; First posted 2012-06-12 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2019-05

CONDITIONS: Infiltrating Bladder Urothelial Carcinoma
Keywords: Bladder cancer; Transitional cell carcinoma; Urothelial cancer; Cisplatin; Cabazitaxel; Chemotherapy; Neo adjuvant chemotherapy
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cabazitaxel + Cisplatin chemotherapy (Experimental): Cabazitaxel 15mg/m2 Intravenous (IV)followed by Cisplatin 70mg/m2 IV on day 1 of each 21 day cycle for 4 cycles
  Interventions: Drug: Cabazitaxel + Cisplatin chemotherapy

INTERVENTIONS:
Drug: Cabazitaxel + Cisplatin chemotherapy — Cabazitaxel 15mg/m2 followed by cisplatin 70mg/m2 given intravenously on day 1 of each 3 weekly cycle for 4 cycles prior to radical cystectomy.
  Other Names: Jevtana

SUMMARY:
26 patients with invasive primary transitional cell carcinoma of the bladder will receive 4 cycles of combination chemotherapy consisting of Cabazitaxel and Cisplatin both given intravenously on day 1 of each 3 weekly cycle prior to radical cystectomy, to evaluate the overall response rate and to determine whether this approach warrants further research of a phase II/III study.Participation in 2 sub studies will also be offered to the participants.

1. Contrast Magnetic resonance imaging (MRI ) scans will be taken at baseline and after cycle 1 and cycle 3.
2. A pilot sub study involving the circulating tumour cell concentration from blood samples taken at baseline, prior to each cycle of chemotherapy and prior to surgery

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically confirmed primary transitional cell carcinoma (TCC) of the urinary bladder
* T2 to T4 disease, N0 M0 determined by computerised tomography (CT) imaging and biopsy or transurethral resection
* Eastern Co-operative Oncology Group (ECOG) Performance status 0 or 1
* Glomerular filtration rate (GFR) ≥60ml/min.
* Written, informed consent

Exclusion Criteria

* ECOG Performance Status ≥ 2
* Lymph node involvement or metastatic disease
* Prior surgery (except transurethral resection of bladder tumour), radiation, che-motherapy, or other anti-cancer therapy within 4 weeks prior to enrolment
* Active Grade ≥2 peripheral neuropathy
* Active secondary cancers
* History of severe hypersensitivity reaction (≥Grade 3) to polysorbate 80 containing drugs
* Other concurrent serious illness or medical conditions
* Inadequate organ function as evidenced by peripheral blood counts at enrolment:
* Electrocardiogram (ECG) evidence of uncontrolled cardiac arrhythmias, angina pectoris, and/or hypertension, history of congestive heart failure, or myocardial infarction within last 6 months.
* Uncontrolled diabetes mellitus.
* Active uncontrolled gastro-oesophageal reflux disease (GORD).
* Active infection requiring systemic antibiotic or anti-fungal medication
* Participation in another clinical trial with any investigational drug within 30 days prior to study enrolment.
* Concurrent or planned treatment with strong inhibitors of cytochrome P450 3A4/5. A 1-week washout period is necessary for patients who are already on these treatments.
* Concurrent or planned treatment with strong inducers of cytochrome P450 3A4/5. A 1-week washout period is necessary for patients who are already on these treatments.
* Contraindications to cisplatin.
* Patient with reproductive potential not implementing an accepted and effective method of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-05; Primary Completion 2017-11 (Actual); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Overall pathological response rate | Histological assessment of radical cystectomy specimen expected to be 15 weeks after commencing study chemotherapy

SECONDARY OUTCOMES:
To record progression free survival | Up to 5 years following radical cystectomy
  From date of registration until the date of first documented progression or date of death from any cause whichever came first.
To assess quality of life | Up to 13 weeks from baseline
  EQ-5D and EORTC QLQC30 and BLM30 will be assessed at baseline and following each cycle of chemotherapy
To record side effects and tolerability of treatment | Up to 13 weeks from baseline
  Common toxicity criteria adverse events (CTC AE ) Version 4.03 will be assessed at baseline and following each cycle of chemotherapy
Overall survival | Up to 5 years following radical cystectomy
  From the date of registration to the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Amit K Bahl, Principal Investigator — University Hospitals Bristol and Weston NHS Foundation Trust
Locations (1):
- Bristol Haematology + Oncology Centre, Horfield Road, Bristol, United Kingdom